CLINICAL TRIAL: NCT03813576
Title: Acceptability and Efficacy of Self-sampling for Cervical Cancer Screening: A Pilot Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2018/00846
Record Dates: First submitted 2019-01-20; First posted 2019-01-23 (Actual); Last update posted 2019-01-23 (Actual); Status verified 2019-01

CONDITIONS: Cervical Cancer; Cervical Dysplasia; Human Papillomavirus Infection
Keywords: screening; cervical cancer; primary prevention; human papillomavirus infection; acceptability; feasibility
MeSH Terms: conditions — Uterine Cervical Neoplasms; Uterine Cervical Dysplasia; Papillomavirus Infections

STUDY DESIGN:
Intervention Model Description: All women will undergo a clinical-collected cervical HPV swab and a self-collected vaginal HPV swab and the results of both swabs compared. The women will be randomised to the sequence of which they undergo the clinical-collected swab first or the self-collected swab first.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All participants (Other): Only 1 arm in the study. All women will undergo both self-collected swab and clinician-collected swab
  Interventions: Diagnostic Test: Self-collected HPV vaginal swab

INTERVENTIONS:
Diagnostic Test: Self-collected HPV vaginal swab — Patients will be instructed on how to collect a vaginal swab on themselves which will then be processed for presence of HPV DNA.

SUMMARY:
In Singapore, the current cervical cancer screening uptake among women in Singapore has remained at low 50% since its introduction in 2004. It has been widely reported that under-screened women have the highest risk of cervical cancer. Self-sampling HPV DNA screening may be a solution to the low uptake rates of local women, particularly among the under-screened population in Singapore. Self-sampling comprises women using a swab to obtain samples from their vagina.

In this study, we are comparing the sensitivity of detecting HPV positive women using HPV DNA test with self-sampling using flocked swab with the current physician sampling method. We also aim to determine acceptability of self-sampling HPV DNA test using flocked swab in cervical cancer screening. Designed as a feasibility study, it will comprise a prospective study of 300 women attending clinics in National University Hospital (NUH) and National Cancer Institute Singapore (NCIS).

DETAILED DESCRIPTION:
Cervical cancer is one of the leading causes of death worldwide. The recognition that cervical cancer is caused by persistent oncogenic HPV virus has caused a considerable paradigm shift in screening and prevention of cervical cancer by the introduction of HPV DNA test and the HPV vaccine. HPV DNA test as an alternative to the current and more traditional cytology only screening has been shown to have higher sensitivity in detecting high grade cervical intraepithelial neoplasia (CIN) to allow for earlier treatment of pre-cancer thus preventing development of cervical cancer in future. Singapore as the rest of the world are in the transition toward the paradigm shift of using HPV DNA test as part of the cervical cancer screening strategy compared to the traditional cytology only screening. However, any cancer screening program to make an impact, an uptake of 70% of more is desired and currently this strategy resulting to the reduction in cervical cancer incidence are only seen in countries adopting an organized cervical cancer screening strategy such as the United Kingdom. Currently, HPV DNA testing has widely been shown to be higher sensitivity to pick up pre-cancer and allow for earlier treatment of pre-cancer. Uptake for cervical cancer screening has remains suboptimal since introduction of the national cervical cancer screening using cytology only method in 2004.

A study published by Jin et.al. in Singapore Medical Journal in 2013 evaluating the progress of cervical cancer screening Singapore (CSS) since its introduction showed that CSS did not make its aim to get 80% uptake for cervical cancer screening for eligible women using cytology only method

Self-sampling in cervical cancer screening

Cervical cancer screening with HPV DNA test is more sensitive than cytology only method to detect pre-cancer cervical cells. It is now well established that cervical cancer screening with HPV DNA test is a much more sensitive method to detect pre-cancer cervical cells compared to cytology only method.

The traditional way of taking a cervical cancer screening involves a physician inserting a speculum into the vagina to visualize the cervix and brushing the surface of the cervix using a cytology brush or spatula. This will collect exfoliated cervical cells to be sent for cytology review to detect any abnormal or pre-cancerous looking cells. Currently HPV DNA test is performed using the same method as taking a pap smear. However, various studies have shown that for HPV DNA test, self-sampling method is a good alternative to physician sampling (Appendix C). Current self-sampling methods in the market are expensive and not cost effective especially if targeting under screeners. There are however, various self-sampling HPV DNA test device in the market. These devices such as the Delphi Screener are expensive and would not be a cost-effective alternative method for women especially in the under screeners in Singapore. Studies have shown that those who do not come for regular cervical cancer screening are usually associated with a lower socioeconomic background. To encourage the under screeners to take up screening, the method should not only be accessible to them but also affordable. The Copan Floq swab has already been used in NUH for Chlamydia testing and it is highly affordable at 3 SGD per swab. Our study would like to determine that using this affordable swab for self-sampling is as sensitive in detecting high risk HPV as a physician sampling method.

There is no local data on the acceptability of self-sampling method using a Floq swab among women in Singapore. The acceptability of self-sampling has been reported to be high among women especially in the western countries. Women in the Asian population in particular Singapore may differ in their acceptability of a self-sampling method compared to a physician sampling method. Self-sampling HPV DNA test will require a woman to insert the cotton swab into the vagina and currently there is no local data to show wether it is an acceptable method for women in Singapore for all ages from 25 to 69 years old. The use of tampons is a much more acceptable method during menstruation in the western country which may influence the acceptability data of self-sampling in the western countries. However, tampon use is not a norm in Asian population including Singapore and may be a factor to influence the acceptability of self-sampling among Singaporean women especially in the older age group.

This study is thus also designed to elucidate this issue. Cervical cancer is a marker of health disparities. Looking to the future, data has shown that failure to go for cervical cancer screening, which is a highly preventable disease, may also be linked to failure of uptake to other screening in a woman. It may also be linked to failure of basic health screening not only for the woman but also for her family. Hence to overcome barriers for cervical cancer screening especially in giving women a reliable alternative option may in future not only help to prevent cervical cancer but also indirectly encourage uptake of other screening such as breast cancer and colorectal screening for her and her family. Our study will attempt to address two questions. 1) Does the self-sampling HPV DNA test as sensitive as the physician sampling HPV DNA test in Singapore? And 2) If Singaporean women have the option of self-sampling, are they more likely to regularly participate in future cervical cancer screening.

STUDY DESIGN

The study is a prospective feasibility study composed of healthy women aged between 30-69 years who are attending clinics in NUH will be identified through the gynaecologist. Ethical approval for this study from the Domain Specific Review Board for O&G is being sought.

Subjects: Three hundred women who meet the inclusion & exclusion below will be invited to participate and complete the consent process. Those that decline will have age, ethnicity, education, work status & reason for declining collected.

Study Visit: Each potential participant will initially see their doctor as clinically intended and offered to participate in the study as identified by each physician in the clinic. Upon agreeing to participate in the study, each participant will be given a study information leaflet and introduced to the research coordination for further explanation of the study and to sign the study consent form. Once consent form is signed, the participant will be given a study self-sampling kit and instructions on how to perform the self-sampling (see Appendix A). The participant performed the self-sampling test in the clinic in a private area and hand over the completed kit to the research coordinator who will label and keep the sample for process.

Post assessment: On completion, the participant will be invited to complete a 10 to 15 minutes questionnaire to assess women's acceptability on self-sampling method. Upon completion of the questionnaire, the participant will be awarded a study token of appreciation prior to leaving the clinic. The participant clinical management will not be affected by the study.

SAMPLE SIZE AND STATISTICAL ANALYSIS

Data collected for this study will be in a password protected Microsoft Excel software. Only the primary investigator and co-investigators will have access to the database for the purpose of data analysis. Sample size was calculated based on the number of women between the ages of 30 and 69 in Singapore's population (as of June 2017). Using a 95% confidence level, it was determined that a sample size of 120 - 150 women would be ideal. The sample size was calculated using G*Power. SPSS will be used to analyze the data collected. Descriptive analyses will be done on the survey data to get demographic data, and to determine participants' perceptions and ratings of the self-sampling methods. Multivariate analyses will be used to determine the sensitivity of the self-sampling method with physician-taken swab as the reference standard.

Data collected will include:

* Patient details: Name and NRIC
* Patient demographics: Age, Race, area code, parity, social economic status
* Reason for HPV DNA test: Primary screening or secondary screening
* Screening results:

  * Physician sampling HPV DNA test
  * Self-sampling HPV DNA test
* Completed questionnaire

Our specific aims are to:

1. To determine the sensitivity of self-sampling method compared to physician sampling method for HPV DNA test in cervical cancer screening
2. To determine acceptability of self-sampling HPV DNA test using flocked swab in cervical cancer screening

The study is designed to give a more accurate local view of the sensitivity of floq swab and acceptability for self-sampling to Singaporean women. Published studies on self-sampling are mainly from the western countries and perception may not be similar for local women. Currently available self-sampling in the market are expensive and thus will not be cost effective if to be introduced to the current Singapore cervical cancer screening program. As Singapore is also moving towards HPV primary screening in the very near future, this study will aid in providing the next step to the screening program by introducing a method that can help to increase uptake of screening in particular in the underscreen population in Singapore.

ELIGIBILITY:
Inclusion criteria: All women aged between 30-69 years who are attending clinics in NUH.

Exclusion criteria:

1. Women who are pregnant
2. Previous total hysterectomy
3. Previous history of cervical cancer
4. Virgin Intacto
5. Negative Pap smear less than 3 years ago.

Ages: 30 Years to 69 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — All participants are female to be applicable for cervical cancer screening
Enrollment: 300 (Estimated)
Dates: Start 2019-03 (Estimated); Primary Completion 2019-08 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity of self-collected HPV swabs | 1 week (time for results of HPV swab to be analysed)
  To determine the sensitivity of self-sampling method compared to physician sampling method for HPV DNA test in cervical cancer screening

SECONDARY OUTCOMES:
Participant acceptability of self-collected HPV swabs | 15 minutes (time for questionnaire to be filled in by participant)
  To determine acceptability of self-sampling HPV DNA test using flocked swab in cervical cancer screening

CONTACTS AND LOCATIONS:
Overall Officials: Ismail Pratt Ida, MBBS, Study Chair — National University Hospital, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Arbyn M, Verdoodt F, Snijders PJ, Verhoef VM, Suonio E, Dillner L, Minozzi S, Bellisario C, Banzi R, Zhao FH, Hillemanns P, Anttila A. Accuracy of human papillomavirus testing on self-collected versus clinician-collected samples: a meta-analysis. Lancet Oncol. 2014 Feb;15(2):172-83. doi: 10.1016/S1470-2045(13)70570-9. Epub 2014 Jan 14. PMID 24433684
- [Result] Petignat P, Faltin DL, Bruchim I, Tramer MR, Franco EL, Coutlee F. Are self-collected samples comparable to physician-collected cervical specimens for human papillomavirus DNA testing? A systematic review and meta-analysis. Gynecol Oncol. 2007 May;105(2):530-5. doi: 10.1016/j.ygyno.2007.01.023. Epub 2007 Feb 28. PMID 17335880
- [Result] Latiff LA, Rahman SA, Wee WY, Dashti S, Andi Asri AA, Unit NH, Siah Li SF, Esfehani AJ, Ahmad S. Assessment of the reliability of a novel self-sampling device for performing cervical sampling in Malaysia. Asian Pac J Cancer Prev. 2015;16(2):559-64. doi: 10.7314/apjcp.2015.16.2.559. PMID 25684487
- [Result] Ketelaars PJW, Bosgraaf RP, Siebers AG, Massuger LFAG, van der Linden JC, Wauters CAP, Rahamat-Langendoen JC, van den Brule AJC, IntHout J, Melchers WJG, Bekkers RLM. High-risk human papillomavirus detection in self-sampling compared to physician-taken smear in a responder population of the Dutch cervical screening: Results of the VERA study. Prev Med. 2017 Aug;101:96-101. doi: 10.1016/j.ypmed.2017.05.021. Epub 2017 Jun 1. PMID 28579497
- [Result] Jin AZ, Louange EC, Chow KY, Fock CW. Evaluation of the National Cervical Cancer Screening Programme in Singapore. Singapore Med J. 2013 Feb;54(2):96-101. doi: 10.11622/smedj.2013032. PMID 23462834
- [Result] Dijkstra MG, Heideman DA, van Kemenade FJ, Hogewoning KJ, Hesselink AT, Verkuijten MC, van Baal WM, Boer GM, Snijders PJ, Meijer CJ. Brush-based self-sampling in combination with GP5+/6+-PCR-based hrHPV testing: high concordance with physician-taken cervical scrapes for HPV genotyping and detection of high-grade CIN. J Clin Virol. 2012 Jun;54(2):147-51. doi: 10.1016/j.jcv.2012.02.022. Epub 2012 Mar 23. PMID 22445557